CLINICAL TRIAL: NCT06980181
Title: Comparison of Graded Motor Imagery and Mirror Therapy in Chronic Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-GCUF-079262
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Speech Disorder; Stroke Rehabilitation; Hypertension
MeSH Terms: conditions — Stroke; Speech Disorders; Hypertension | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Investigator
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Motor Imagery (Experimental): GMI uses visual cues and mental exercises to retain the brain in steps.
  Interventions: Other: Graded Motor Imagery
- Mirror Therapy (Active Comparator): Mirror Therapy uses a mirror to make the brain think the weak side is moving
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Graded Motor Imagery — Graded Motor Imagery typically 1 to 3 times per day for 5 to 10 minutes for each phase. No physical movement at first only cognitive task, mental rehearsal and visual motor.
  Arms: Graded Motor Imagery
Other: Mirror Therapy — Mirror Therapy typically involves 1 to 3 sessions per day for 10 to 15 minutes gradually increases as tolerated.Visual and motor training using a mirror placed at the midline.
  Arms: Mirror Therapy

SUMMARY:
The study is conducted to assess whether the GMI or MT reduce the level of spasticity. Also to compare the level of independence in GMI and MT in the chronic stroke patients.

DETAILED DESCRIPTION:
A stroke is a medical condition that occurs when inadequate blood flow to a part of the brain leads to cell death. There are two primary types of strokes: ischemic, caused by reduced blood flow, and hemorrhagic, caused by bleeding. Both types result in impaired brain function in the affected areas.

A systemic review was conducted on the effectiveness of mirror therapy on lower extremities, stal and walk in early stage and long term stroke. Results shown better results with using mirror the than control group.

Non-randomized controlled trial study was conducted on stroke patients treated by graded n imagery. It consisted of 28 subjects and the experimental group included 14 and other 14 included in the control group. Graded motor imagery showed better results than the convent therapy as 10 patients showed better outcomes in the intervention group and only 4 patients sho improvement in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age:45 to 65 years
* First ever unilateral stroke and over 3 months since onset.
* Both ischemic and hemorrhagic stroke individuals were included.

Exclusion Criteria

* Patients suffering from psychological problems.
* Visual Impairments.
* Fractures.
* Any other Neurological disorder
* Inflammatory joint diseases
* Medical instability e.g Uncontrolled HTN
* Any systemic disease

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 4 weeks
  Changes from baseline Modified Ashworth SCale is a clinical tool used to measure the spasticity.It comprises 4 grades.0 No increase in muscle tone, 1 Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM), 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM, 2 More marked increase in muscle tone through most of the ROM, but affected parts) easily moved, 3 Considerable increase in muscle tone, passive movement difficult, 4 Affected parts rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Usman Iqbal Janjua, Phd, Principal Investigator — Elite College of Management Sciences
Locations (1):
- Paraplegic Center, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandhi DB, Sterba A, Khatter H, Pandian JD. Mirror Therapy in Stroke Rehabilitation: Current Perspectives. Ther Clin Risk Manag. 2020 Feb 7;16:75-85. doi: 10.2147/TCRM.S206883. eCollection 2020. PMID 32103968
- [Background] Gallanagh S, Quinn TJ, Alexander J, Walters MR. Physical activity in the prevention and treatment of stroke. ISRN Neurol. 2011;2011:953818. doi: 10.5402/2011/953818. Epub 2011 Oct 1. PMID 22389836